CLINICAL TRIAL: NCT02942368
Title: Adaptive Transcranial Direct Current Stimulation as an Adjunctive Therapy for Treatment-Resistant Major Depressive Disorder
Brief Title: Adaptive tDCS for Treatment-Resistant MDD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6610-201610133
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Treatment-Resistant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Masking Description: Outcomes assessors are blinded and unaware of the specifics of the study (although only a single arm, blinded raters do not know this).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- tDCS (Experimental): Patients will receive transcranial direct current stimulation using an adaptive protocol allowing for doses of 0 to 4 mA during the course of the treatment, with twenty 20-minute sessions over the course of 4 to 6 weeks. Treatments will take place daily, 5 days per week.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Transcranial direct current stimulation with placement of the anode over the F3 region of the scalp and the cathode over the right supraorbital region.

SUMMARY:
This pilot study aims to investigate the potential role of transcranial direct current stimulation (tDCS) in the treatment of treatment-resistant major depressive disorder (MDD). tDCS is a noninvasive brain stimulation technique which has been utilized for the treatment of major depression in several studies, both as a primary and adjunctive treatment. The treatment will be administered under the supervision of a physician with experience in administering the treatment and monitoring for complications. This will be a prospective "adaptive tDCS stimulation" open label research study. Participants will receive 20 minute sessions of up to 4 milliamps (mA) transcutaneous electrical stimulation sessions over 4 to 6 weeks. Building on the theory that greater current "dose" may be a significant factor in determining efficacy, this study aims to determine whether higher tDCS current doses lead to greater improvements in depressive symptoms in this population of patients with treatment-resistant major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Adults age 18 to 65
2. History of major depressive disorder with current depressive symptoms, as defined by DSM-IV criteria
3. Baseline score of Hamilton Depression Rating Scale 17-item (HDRS-17) score of 17 or higher
4. Failure of at least 3 prior lifetime antidepressant trials
5. Good command of the English language

Exclusion Criteria:

1. Lifetime history of the following, defined by DSM-IV criteria per study physician:

   1. Moderate or severe substance use disorder in the past 6 months with the exception of nicotine use disorder
   2. Dementia or major neurocognitive disorder
   3. Schizophrenia spectrum disorders
   4. Autism spectrum disorder
   5. Depression which has failed to respond to ECT, with treatment failure as determined by evaluating physician
   6. Failure of greater than 6 antidepressant trials in the current depressive episode
2. Current evidence of the following, defined by present symptomology as per study physician:

   1. Active psychotic symptoms
   2. Bipolar disorder with a current manic, hypomanic, or mixed episode as defined by DSM-IV criteria
   3. Depression secondary to a general medical illness
   4. Dysphoria better explained by a personality disorder
   5. Dysphoria associated with a primary anxiety disorder or PTSD
   6. Active suicidal intention (inability to contract for safety)
   7. Any change in psychotropic medication within 30 days of the initiation of tDCS
   8. History of neurological disorders (e.g., epilepsy) and/or off any treatment medication for a neurological disorder for minimum 3 years (36 months)
   9. Any open wounds (e.g., blisters, burns including sun burns, cuts or irritation) under or near the scalp regions where electrodes are placed
   10. Metal implants (e.g., Deep Brain Stimulator, Vagus Nerve Stimulator)
   11. Any skin disorders (e.g., eczema, severe rashes, sensitive skin, any communicable skin disorder or treatment for a communicable skin disorder in the past 12 months) or other skin defects which compromise the integrity of the skin at or near stimulation locations (where electrodes are placed)
   12. Any history of head injury resulting in unconsciousness for more than 5 minutes (e.g., head trauma, brain surgery)
   13. Metallic face or scalp tattoos
   14. Any chronic headaches or migraines (occurring for consecutive days and are longer than an hour)
   15. If a participant has a change in the rate or severity of head pressure, headache, or migraine in the past two weeks, they will also be excluded as per study clinician as we are not aiming to assess the treatment of headache with tDCS
   16. Any personal history of seizures.
3. Currently pregnant or lactating, as determined in part from urine pregnancy test at Screening/Baseline appointment and medical history.
4. Any other factor that in the investigators' judgment may affect patient safety or compliance (e.g. distance greater than 100 miles from clinic)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2017-04-14 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in depressive symptoms as measured by mean change in the Montgomery-Åsberg Depression Rating Scale (MADRS) score from baseline to end of the study. | Measurements at week 0, week 2, week 4, week 5 and week 6

CONTACTS AND LOCATIONS:
Overall Officials: Charles Conway, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in Saint Louis, St Louis, Missouri, United States